CLINICAL TRIAL: NCT01319526
Title: Quantification of HIV-1 Reservoirs in HIV-Positive Persons Receiving Response-Adapted Therapy for Stage III-IV Hodgkin Lymphoma: A Companion Protocol to SWOG Protocol S0816 (AMC-073)
Brief Title: Biomarkers in Blood Samples From Patients With HIV Infection and Stage III or Stage IV Hodgkin Lymphoma Undergoing Chemotherapy
Status: Terminated | Type: Observational
Why Stopped: Parent protocol (SWOG S0816 / AMC-073) discontinued
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: AMC-079; CDR0000690149 (Other: NCI)
Record Dates: First submitted 2010-12-18; First posted 2011-03-21 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Lymphoma; Nonneoplastic Condition
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; HIV infection
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PBMC
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA analysis
Genetic: RNA analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory from patients undergoing treatment with HIV infection and Hodgkin lymphoma may help doctors learn more about the effects of therapy on HIV.

PURPOSE: This research study is studying biomarkers in blood samples from patients with HIV infection and stage III or stage IV Hodgkin lymphoma undergoing chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To quantify HIV-1 persistence in prospectively collected samples from patients on suppressive antiretroviral therapy undergoing chemotherapy for Hodgkin lymphoma.

OUTLINE: This is a multicenter study.

Blood samples are collected before, during, and after treatment for lymphoma for HIV-1 RNA levels using standard and single copy assays and HIV-1 DNA quantification (peripheral blood mononuclear cells).

After completion of treatment, patients are followed up periodically for up to 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* HIV-1 infection, as documented by a rapid HIV test or any FDA-approved HIV-1 enzyme or chemiluminescence immunoassay (E/CIA) test kit and confirmed by western blot at any time prior to study entry

  * Documentation may be serologic (positive ELISA and positive western blot), or other federally approved licensed HIV diagnostic test
  * Prior documentation of HIV seropositivity is acceptable
* Diagnosis of untreated Hodgkin lymphoma and participation in the parent protocol SWOG-S0816, "A Phase II Trial of Response Adapted Therapy of Stage III-IV Hodgkin Lymphoma Using Early Interim FDG-PET Imaging."

PATIENT CHARACTERISTICS:

* No psychosocial conditions that would prevent study compliance and follow-up, as determined by the principal investigator
* Willing to provide serial blood samples

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical trial participants (subjects who are participating in parent protocol S0816 and provide informed consent for participation in this substudy).
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in viral load from baseline to each subsequent time point | Baseline, after each cycle of treatment, restaging, treatment completion, year 1, year 2, study discontinuation
  Time frame for outcome measures dependent on study calendar for parent protocol, S0816, which varies by subject's PET scan status.

CONTACTS AND LOCATIONS:
Overall Officials: John W. Mellors, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts